CLINICAL TRIAL: NCT00000680
Title: A Phase I Study of Autologous, Activated CD8(+) Lymphocytes Expanded In Vitro and Infused With or Without Recombinant Interleukin-2 to Patients With AIDS or Severe ARC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Applied Immunesciences (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 080; 11055 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes, Suppressor-Effector; Indium Radioisotopes; Leukapheresis; Interleukin-2; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Immunization, Passive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; aldesleukin

INTERVENTIONS:
Drug: Zidovudine
Drug: Aldesleukin

SUMMARY:
1) To determine whether it is possible to remove and culture (increase in number and activate) in the laboratory, CD8(+) lymphocytes (white blood cells) from HIV-infected patients receiving zidovudine (AZT); 2) To determine the toxicity of returning to the patients intravenously the expanded and activated autologous cells (given to the patient from whom they were taken), with and without giving the patients recombinant interleukin-2 ( aldesleukin; IL-2 ) at the same time; 3) To radiolabel (mark) the CD8(+) lymphocytes with Indium 111, and then scan the patients to determine the distribution of the CD8(+) lymphocytes in those who are and are not given IL-2 infusions; 4) To determine the toxicity of IL-2 given at the same time with autologous CD8(+) lymphocytes; 5) To measure changes in the immunology of the subjects following these treatments.

CD8(+) cells are suppressor/killer lymphocyte cells that act to limit replication of viruses. It is hoped that the reinfusion of activated autologous CD8(+) cells into patients with AIDS will help to control opportunistic infections such as cytomegalovirus and toxoplasmosis (two of the leading causes of sickness and death in AIDS patients). This treatment may also stop the HIV virus from replicating (reproducing itself) in the AIDS patient. Further activation of these cells, once infused, may be necessary. It is hoped that IL-2 will stimulate the patient's immune system against the AIDS virus along with the activated CD8(+) cells. Thus, IL-2 will be given, and its effects studied.

DETAILED DESCRIPTION:
CD8(+) cells are suppressor/killer lymphocyte cells that act to limit replication of viruses. It is hoped that the reinfusion of activated autologous CD8(+) cells into patients with AIDS will help to control opportunistic infections such as cytomegalovirus and toxoplasmosis (two of the leading causes of sickness and death in AIDS patients). This treatment may also stop the HIV virus from replicating (reproducing itself) in the AIDS patient. Further activation of these cells, once infused, may be necessary. It is hoped that IL-2 will stimulate the patient's immune system against the AIDS virus along with the activated CD8(+) cells. Thus, IL-2 will be given, and its effects studied.

AMENDED: 09/28/90 The CD8 lymphocytes are grown in vitro for 21 days before infusion. Leukapheresis and infusion continue every 21 days for 3 infusions with the last infusion during week 16. During weeks 13 and 16, indium 111 radio labelled cells are injected to permit determination of the distribution and pharmacokinetics of the infused cells. At week 16, IL-2 is administered concurrently with Indium 111 labelled cells and the CD8+ lymphocytes - delivered by continuous infusion over 5 days following cell infusion. Patients are followed at the clinic 1 week prior to scheduled infusions, during infusion weeks and then every 2 weeks to week 21 and at week 27. Original design: Patients undergo leukapheresis every 2 weeks for a total of 6 times during the initial phase of the study. During this procedure, a catheter is placed in an arm vein, and the blood flows through a machine which separates the lymphocytes from the other blood components. The blood is then returned to the patient's body through the catheter. Less than 10 percent of the lymphocytes in the blood are removed during the process. The CD8(+) cells taken from the patient are cultured in the laboratory until they increase 10- to 1000-fold. These cells are then infused back into the patient from whom they were taken. The first two patients are admitted for 24 hours at the time of each infusion. In the absence of severe side effects, the subsequent four patients are infused at the clinic. Patients are admitted for 5 days for continuous infusion of IL-2 in week 13.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Zidovudine (AZT) during treatment and for 20 weeks after the last infusion unless medically contraindicated.
* Allowed:
* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Oral antibiotics for PCP prophylaxis if hematologically stable on that regimen for at least 30 days prior to study entry.

Patients must have the following:

* Positive HIV antibody test by federally licensed ELISA.
* Positive HIV culture or plasma p24 antigen.
* CDC Group IV severe AIDS-related complex (ARC) or AIDS.
* Must have been on zidovudine (AZT) at least 6 weeks prior to infusion and agree to continue this medication during the study and for 20 weeks after the last infusion unless medically contraindicated.
* Allowed:
* Kaposi's sarcoma.

Exclusion Criteria

Co-existing Condition:

AMENDED:

* Pulmonary diseases that require treatment.
* AMENDED:
* Significant central nervous system disease including AIDS dementia, psychiatric disabilities, or seizure disorders.
* AMENDED:
* Symptomatic HIV CNS infections or symptoms compatible with HIV encephalopathy.
* Original design:
* Patients with the following conditions or symptoms are excluded:
* Active bacterial or opportunistic infection that requires treatment.
* Neoplasms not specifically allowed, basal cell carcinoma of the skin, or in-situ carcinoma of the cervix.
* Clinically significant cardiac (= or > class II, New York Heart Association) or peripheral vascular disease that requires treatment.
* Hemorrhagic diathesis including hemophilia or active bleeding disorder.

Concurrent Medication:

Excluded:

* Antineoplastic therapy.
* Medication required for treatment of active cardiac disease.
* Cardiac glycosides.
* Antiarrhythmics.
* Antianginal agents.
* Anticoagulants.
* Thrombolytic agents.
* Vasodilators.
* Excluded within 30 days of study entry:
* Antiretroviral agents not specifically allowed.
* Corticosteroids.
* Acyclovir.
* Excluded within 60 days of study entry:
* Biological response modifiers.

Patients with the following are excluded:

* Unable to give properly informed consent by reason of impaired mentation.
* Diseases and conditions specified elsewhere in the protocol.

Required:

* Zidovudine (AZT) for at least 6 weeks prior to infusion.

Risk Behavior: Excluded:

* Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Study Completion 1993-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Ho, Study Chair; R Herberman, Study Chair; J Armstrong, Study Chair
Locations (1):
- Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Torpey D 3rd, Huang XL, Armstrong J, Ho M, Whiteside T, McMahon D, Pazin G, Heberman R, Gupta P, Tripoli C, et al. Effects of adoptive immunotherapy with autologous CD8+ T lymphocytes on immunologic parameters: lymphocyte subsets and cytotoxic activity. Clin Immunol Immunopathol. 1993 Sep;68(3):263-72. doi: 10.1006/clin.1993.1127. PMID 8370181
- [Background] Ho M, Armstrong J, McMahon D, Pazin G, Huang XL, Rinaldo C, Whiteside T, Tripoli C, Levine G, Moody D, et al. A phase 1 study of adoptive transfer of autologous CD8+ T lymphocytes in patients with acquired immunodeficiency syndrome (AIDS)-related complex or AIDS. Blood. 1993 Apr 15;81(8):2093-101. PMID 8471768
- [Background] Ho M, et al. Phase I study of in vitro purified and expanded autologous CD8(+) lymphocytes infused into patients with advanced ARC or AIDS (ACTG 080). Int Conf AIDS. 1991 Jun 16-21;7(2):77 (abstract no THB83)
- [Background] Armstrong JA, Ho M, Herberman R, Elder E, Ferbas J, McMahon D, Gupta P, Rinaldo C, Whiteside T. A phase I study of autologous, activated CD8(+) lymphocytes expanded in vitro infused into patients with advanced ARC or AIDS (ACTG 080). Int Conf AIDS. 1990 Jun 20-23;6(3):208 (abstract no SB491)